CLINICAL TRIAL: NCT00002748
Title: Phase I Study of Cytokine-Gene Modified Autologous or Partially Matched Allogeneic Neuroblastoma Cells for Treatment of Relapsed/Refractory Neuroblastoma
Brief Title: Gene Therapy in Treating Children With Refractory or Recurrent Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064681; U01CA058211 (NIH); P30CA021765 (NIH); SJCRH-CYGENE; SJCRH-CYGNE2; NCI-H96-0005
Record Dates: First submitted 1999-11-01; First posted 2004-01-22 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Interleukin-2

INTERVENTIONS:
Biological: gene-modified tumor cell vaccine therapy
Biological: interleukin-2 gene

SUMMARY:
RATIONALE: Inserting the gene for interleukin-2 into a person's neuroblastoma cells may make the body build an immune response and kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of using interleukin-2 gene-modified neuroblastoma cells in treating children who have refractory or recurrent neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety in children of recurrent neuroblastoma of two weekly subcutaneous injections of autologous, or partially HLA-matched allogeneic, neuroblastoma cells that have been modified by insertion of the interleukin-2 gene introduced by a retroviral vector. II. Determine whether multiple histocompatibility-restricted or unrestricted antitumor immune responses are induced by this treatment and the cell dose required to produce these effects. III. Obtain preliminary data on the antitumor effects of this regimen.

OUTLINE: Autologous or partially HLA-matched allogeneic neuroblastoma cells are transduced with a human gene for interleukin-2 production. Patients receive subcutaneous injections of the gene-modified cells on days 1 and 8, with the second injection containing 10 times more cells than the first injection. After a 3-4 week rest, stable and responding patients may receive additional weekly injections at the second dose. Cohorts of 3-6 patients will be entered at increasing cell doses until the maximum tolerated dose is estimated. Multiple injection sites may be used at the higher cell-dose levels. Patients are followed every week for 6 weeks, every other week for 6 weeks, and monthly for 1 year. Additional visits may be required as clinically indicated.

PROJECTED ACCRUAL: Approximately 12 patients each will be entered into the autologous and the partially HLA-matched allogeneic tumor cell treatment groups. Accrual is expected to require 4 years for the autologous tumor cell group and 2 years for the partially HLA-matched allogenic tumor cell group.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven high risk neuroblastoma at the completion of planned primary therapy No rapidly progressing disease Allogeneic transduced cell line available Demonstrated production of at least 150 picograms of interleukin-2 per 10 to the 6th cells per day

PATIENT CHARACTERISTICS: Age: Under 21 at diagnosis Performance status: ECOG 0-2 Life expectancy: At least 8 weeks Hematopoietic: (unless marrow replaced by tumor) Absolute neutrophil count greater than 500/mm3 Platelet count greater than 50,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL AST no greater than 2 times normal PT normal Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 80 mL/min Urinalysis normal Metabolic: Electrolytes (including calcium, phosphate) normal Glucose normal Weight greater than 10th percentile for age Albumin greater than 3 g/dL Other: No active infection HIV negative Not pregnant or nursing

PRIOR CONCURRENT THERAPY: See Disease Characteristics Recovered from prior chemotherapy No concurrent antibiotics except prophylactic trimethoprim/sulfamethoxazole No concurrent drugs other than analgesics

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 1991-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hale, MD, Study Chair — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org